CLINICAL TRIAL: NCT04315272
Title: Gut and Azithromycin Mechanisms in Infants and Children II
Acronym: GAMINII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPP1187628-D
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Individually randomized placebo-controlled trial of azithromycin vs. placebo to establish the efficacy and safety of azithromycin.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Active Comparator): A single dose of azithromycin will be administered to children between the ages of 8 days and 59 months old.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): A single dose of placebo will be administered to children between the ages of 8 days and 59 months old.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Zithromax® for oral suspension is supplied in bottles containing azithromycin dehydrate powder equivalent to 1200mg per bottle and the following inactive ingredients: sucrose; tribasic anhydrous sodium phosphate; hydroxypropyl cellulose; xanthan gum; FD&C Red #40; and flavoring including spray dried artificial cherry, crème de vanilla, and banana. After constitution, a 5mL suspension contains 200mg of azithromycin.
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Childhood mortality is decreasing worldwide. However, many sub-Saharan countries still have high children under 5 mortality rates. The MORDOR trial in Niger, Tanzania, and Malawi demonstrated a near 14% decrease in all-cause child mortality following biannual azithromycin in children 1-59 months. Current trials in Burkina aim to replicate these results from the MORDOR study with mass azithromycin treatment.

The investigators conducted an individually randomized placebo-controlled trial in Burkina Faso called the Gut and Azithromycin Mechanisms in Infants and Neonates Trial (GAMIN: NCT03676751) to evaluate the effect of a single dose of azithromycin (20 mg/kg) on potential mediators of the effect of azithromycin on all-cause mortality and to evaluate changes in the gut microbiome longitudinally (results pending). Here, the investigators propose to conduct an expansion of the original GAMIN trial. In GAMIN II, the investigators will evaluate 450 additional 1-59 month old children longitudinally for 6 months with a focus on stool collection and malaria status.

Objectives:

1. To determine the effect of a single dose of azithromycin for children aged 8 days-59 months on malaria. The investigators hypothesize that a single dose of azithromycin will result in a reduced malaria status within the treatment group compared to the placebo group after a 14 day period within children ages 8 days-59 months.

The study will be conducted in Nouna Town in northwestern Burkina Faso.

DETAILED DESCRIPTION:
The investigators' previous MORDOR I research demonstrated a significant reduction in all-cause child mortality after biannual mass azithromycin distribution. In three sub-Saharan Africa countries, (including Niger, Tanzania, and Malawi) mass azithromycin treatment over 2 years resulted in a 14% reduction in child mortality. Moreover, 1 in 5-6 deaths were shown to be averted within Niger alone1. Similar findings were demonstrated in a previous study for trachoma control in Ethiopia with mass azithromycin distribution. This study in rural Ethiopia noted a nearly 50% decrease in all-cause childhood mortality5. However, neither of these studies evaluated the longitudinal impact azithromycin has on the gut microbiome. The MORDOR II trial in Burkina Faso will further evaluate the efficacy of biannual azithromycin treatment. The under-5 child mortality rate in Burkina Faso is approximately 110 per 1,000 live births. Major causes of child mortality in this area are infectious mostly due to malaria, diarrhea, and upper respiratory tract infections. In addition, malnutrition contributes to a high burden of child mortality and morbidity within this region as well. By treating underlying conditions, the use of routine antibiotic treatment could reduce diverse health outcomes leading to morbidity and mortality. The investigative team proposes to conduct this study alongside the MORDOR II trial in the town of Nouna where a majority of childhood deaths are attributable to infectious causes and malnutrition.

The World Health Organization is considering adopting the presumptive use of azithromycin and other antibiotics as a recommendation to reduce childhood mortality in areas with a high infectious disease burden. Many questions remain unanswered surrounding the use of mass antibiotic treatment in areas with high child morbidity and mortality. This study will add to the current knowledge of mass azithromycin distribution from our previous MORDOR I research. The investigators propose to evaluate how azithromycin will impact childhood growth and to assess the changes that occur in the intestinal microbiome following a single dose of azithromycin treatment. The goal is to contribute more scientific literature that could assist future guidelines regarding antibiotic use.

The role of antibiotics on the gut microflora is unclear. Longitudinal studies have been recommended to further investigate the role of antibiotics on the microbiome. The investigators propose a longitudinal study designed to improve our knowledge about the changes in the intestinal microbiome following the course of a single dose of antibiotic in a setting with high childhood mortality and morbidity. More specifically, the investigators propose to follow 450 children for a 6-month time period that are between the ages of 8 days old and 59 months old. Children in this age bracket are at the highest risk for mortality from infectious causes, and furthermore, they are at the highest risk for malnutrition. This group of children would receive the greatest benefit from this intervention. The causal changes in the microbiome are vastly understudied in regards to changes in the gut microbiome following a course of antibiotics. Additionally, this study will provide valuable data on the effect of azithromycin for malaria status within 2 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 days and 59 months old
* Primary residence within catchment area of study site
* Available for full 6 month study
* No known allergy to macrolides/azalides
* Appropriate written informed consent from at least one parent or guardian
* Able to feed orally

Exclusion Criteria:

* <8 days old or >59 months
* Primary residence outside catchment area of study site
* Not available for full 6 month study
* Known allergy to macrolides/azalides
* No written informed consent from at least one parent or guardian
* Unable to feed orally

Ages: 8 Days to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catie Oldenburg, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de Recherche en santé de nouna, Nouna, Boucle du Mouhoun, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brogdon J, Dah C, Sie A, Bountogo M, Coulibaly B, Kouanda I, Ouattara M, Compaore G, Nebie E, Seynou M, Lebas E, Nyatigo F, Hu H, Arnold BF, Lietman TM, Oldenburg CE. Malaria positivity following a single oral dose of azithromycin among children in Burkina Faso: a randomized controlled trial. BMC Infect Dis. 2022 Mar 25;22(1):285. doi: 10.1186/s12879-022-07296-4. PMID 35337289

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: 8 days to 59 months old were randomized to a single oral dose of azithromycin (20 mg/kg) Azithromycin: Zithromax® for oral suspension is supplied in bottles containing azithromycin dehydrate powder equivalent to 1200mg per bottle and the following inactive ingredients: sucrose; tribasic anhydrous sodium phosphate; hydroxypropyl cellulose; xanthan gum; FD&C Red #40; and flavoring including spray dried artificial cherry, crème de vanilla, and banana. After constitution, a 5mL suspension contains 200mg of azithromycin.
- Placebo: A single dose of placebo will be administered to children between the ages of 8 days and 59 months old.
  Placebo: Oral suspension of placebo for azithromycin
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 221 | 228
Completed | 220 | 227
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 221 | 228 | 449
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 32 [21 to 44] | 32.5 [22 to 44.5] | 32 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 110 | 217
  Male | 114 | 118 | 232
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 221 | 228 | 449
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Burkina Faso | 221 | 228 | 449
Mother's age, years [Median (Inter-Quartile Range); unit: years] | 26 [23 to 31] | 27 [23 to 32] | 27 [23 to 32]
Currently breastfeeding [Count of Participants; unit: Participants] | 64 | 51 | 115
Mother is literate [Count of Participants; unit: Participants] | 92 | 97 | 189

OUTCOME MEASURES:

1. Primary Outcome: Malaria Status
Description: A rapid diagnostic test will be administered to all children to determine malaria status
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 220 | 227
Participants | 18 | 16

2. Secondary Outcome: Clinical Malaria
Description: Clinical malaria will be defined by a positive rapid diagnostic test and fever.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 220 | 227
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 14 days following azithromycin or placebo treatment
Description: We report adverse events and clinic visits during the 2-week period immediately after treatment to better understand the safety and short-term impact of azithromycin compared with placebo in young children.
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/227
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/227
Other Adverse Events (participants affected / at risk) | 20/220 | 32/227
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=220) | Placebo (N=227)
Fever (General disorders) | 8 | 19
Abdominal pain (General disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 11 | 18
Vomiting (Gastrointestinal disorders) | 6 | 14
Constipation (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04315272/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT04315272/SAP_001.pdf